CLINICAL TRIAL: NCT06925139
Title: Efficacy of Non-Ablative Radiofrequency on Vaginal and Sexual Health in Postmenopausal Women: a Randomized Clinical Trial
Brief Title: Efficacy of Non-Ablative Radiofrequency on Vaginal and Sexual Health in Postmenopausal Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEN_RF_01
Record Dates: First submitted 2024-06-05; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Genitourinary Syndrome of Menopause; Vaginal Health; Sexual Dysfunction
Keywords: Non-ablative radiofrequency; Vaginal Health; Sexual Health; Postmenopause; Genitourinary Syndrome of Menopause; Sexual Dysfunction; Women's Health
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: This study is a double-blind, randomized clinical trial with two parallel groups. Participants are randomly assigned to one of two groups: the treatment group receiving non-ablative monopolar radiofrequency and the placebo group receiving a sham procedure. Both participants and researchers are blinded to group assignments to ensure unbiased results. The study includes six treatment sessions for each participant, with evaluations conducted at baseline, at the end of the treatment period, and three months post-treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this double-blind, randomized clinical trial, participants, investigators analyzing the results, and outcomes assessors are all blinded to the group assignments. This ensures unbiased administration of treatments, unbiased data collection, and unbiased assessment of both primary and secondary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): 6 treatment sessions of non-ablative radiofrequency, with a frequency of 1 session per week. The following protocol will be followed: Preparation (5 minutes): Resistive monopolar electrode applied to vulvar area with gradual heating (sensation 4-5/10).
  Main Phase (15 minutes): Intracavitary capacitive electrode used to reach and maintain 40-42°C for at least 10 minutes.
  Final Phase (5 minutes): Repeat resistive electrode application with subthermal effect (sensation 3-4/10).
  Interventions: Device: Non-ablative monopolar radiofrequency treatment
- Placebo Group (Sham Comparator): Participants in this group will receive the same treatment protocol, but without the application of heat.
  Interventions: Device: Non-ablative monopolar radiofrequency treatment

INTERVENTIONS:
Device: Non-ablative monopolar radiofrequency treatment — Protocol for the experimental group:
  Tissue preparation phase: 5 minutes with the circular resistive monopolar electrode, applying slow circular or semicircular movements in the perineal area. The temperature will be gradually increased based on the patient's temperature perception, ensuring it remains comfortable (approximately 5 out of 10).
  Main phase: 10 minutes using the intracavitary capacitive electrode connected to the PLUMA handle, lightly resting it on the tissues and continuously moving the electrode. The temperature should reach 40-42°C in the tissue and be maintained for at least 10 minutes.
  Final phase: 5 minutes with the circular resistive monopolar electrode, applying it similarly to the preparatory phase, with a subthermal effect, reaching a self-reported thermal sensation of 3 to 4 out of 10.
  Protocol for the sham group: this group will receive the same treatment protocol that treatment group, but without the application of heat.

SUMMARY:
This study will test if non-ablative monopolar radiofrequency can help improve vaginal tissue and reduce symptoms of Genitourinary Syndrome of Menopause (GSM) in postmenopausal women. The study is a double-blind, randomized clinical trial. The study will examine the impact of the treatment on sexual function, vaginal health, and quality of life over an extended period. There will be two groups in the study: one will receive the non-ablative monopolar radiofrequency treatment, and the other will receive the placebo treatment. Participants will have six treatment sessions and will be checked at the start, end, and three months post-treatment.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of non-ablative monopolar radiofrequency (RF) treatment in improving vaginal tissue regeneration and alleviating symptoms of Genitourinary Syndrome of Menopause (GSM) in postmenopausal women. This double-blind, randomized clinical trial will include two groups: one receiving the active RF treatment and the other receiving a placebo treatment. The study will include six treatment sessions for each participant, with evaluations conducted at baseline, at the end of the treatment period, and three months post-treatment.

Participants will be postmenopausal women who have experienced more than one year of amenorrhea and exhibit symptoms of GSM, such as vaginal dryness, irritation, and sexual dysfunction. The primary outcome measures will include improvements in vaginal health assessed through clinical examination and patient-reported outcomes related to sexual function and quality of life.

Secondary outcome measures will involve the analysis of vaginal pH, the maturation index of vaginal epithelial cells, and any adverse events reported during the study. The intervention involves the use of a non-ablative monopolar RF device applied intracavitarily. The placebo group will undergo the same procedure without the active RF component.

The study is conducted in accordance with ethical standards and has been reviewed and approved by the Ethics Committee for Clinical Research with Medicines of the City of Toledo. Data will be collected and analyzed to determine the effectiveness of the treatment in comparison to the placebo, and results will contribute to the understanding of non-ablative RF treatments in menopausal health.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65 years.
* Postmenopausal women (defined as no menstrual period for at least 12 months).
* Experiencing symptoms of Genitourinary Syndrome of Menopause (GSM), such as vaginal dryness, irritation, or discomfort.
* Experiencing discomfort or complaints during vaginal penetration. Engaging in sexual activity (at least once a month).
* Willing to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Presenting with active vaginal infections.
* Presence of neurological, neoplastic, or sexually transmitted diseases.
* Presenting with vulvodynia or vaginismus.
* Prolapse grade 2 or higher.
* Presenting with altered sensitivity in the pelvic area.
* Being a pacemaker carrier or having any device that contains batteries.
* Hormonal treatment with estrogens in the last 3 months.
* History of radiotherapy in the pelvic area.
* Recent pelvic surgery (within the last 6 months).
* Being on anticoagulant treatment.
* Having undergone laser treatment in the pelvic area or ablative vaginal rejuvenation in the last 6 months.
* Cognitive impairment that prevents answering the questionnaires.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified females who are biologically female and postmenopausal.
Enrollment: 58 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in Female Sexual Function Index (FSFI) | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Multidimensional questionnaire evaluates sexual function over the past 4 weeks. The total score ranges from 2.0 (severe dysfunction) to 36.0 (no dysfunction). Sexual dysfunction was defined as a score equal to or below 26.55
Change in Vaginal Health Index (VHI) | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  A tool that evaluates five parameters: vaginal elasticity, vaginal secretion (type and consistency), pH, mucosal epithelial integrity, and vaginal moisture. Each parameter was scored on a scale from 1 (most unfavorable condition) to 5 (optimal condition), with a maximum possible score of 25 points. In cases where the score was below 15, the vagina was considered atrophic.

SECONDARY OUTCOMES:
Change in sexual desire | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Female Sexual Function Index in individual domain of sexual desire. Score from 1,2 (worst) to 6 (best)
Change in sexual arousal | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Female Sexual Function Index in individual domain of sexual arousal. Score from 0 (worst) to 6 (best)
Change in sexual lubrication | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Female Sexual Function Index in individual domain of sexual lubrication. Score from 1,2 (worst) to 6 (best)
Change in sexual orgasm | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Female Sexual Function Index in individual domain of sexual orgasm. Score from 0 (worst) to 6 (best)
Change in sexual satisfaction | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Female Sexual Function Index in individual domain of sexual satisfaction. Score from 0.8 (worst) to 6 (best)
Change in sexual pain | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Female Sexual Function Index in individual domain of sexual pain. Score from 0 (the worst possible pain) to 6 (no pain).
Change in vaginal Elasticity | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Vaginal Health Index in individual domain of vaginal elasticity. Score from 1 (most unfavorable condition) to 5 (optimal condition)
Change in Vaginal secretion | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Vaginal Health Index in individual domain of vaginal secretion. Score from 1 (most unfavorable condition) to 5 (optimal condition)
Change in vaginal pH | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Vaginal Health Index in individual domain of vaginal pH. Score from 1 (most unfavorable condition) to 5 (optimal condition)
Change in vaginal Ephitelial integrity | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Vaginal Health Index in individual domain of vaginal ephitelial integrity. Score from 1 (most unfavorable condition) to 5 (optimal condition)
Change in vaginal Moisture | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Assessed by Vaginal Health Index in individual domain of vaginal moisture. Score from 1 (most unfavorable condition) to 5 (optimal condition)
Change in Vaginal Maturity Index | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  The proportion of parabasal, intermediate, and superficial cells in each 100 cells counted on a smear of the upper two-thirds of the vagina.
Change in Status Estrogen | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  This index will be calculated using Meisels' formula: (% intermediate cells × 0.5 + % superficial cells).
Change in Vaginal Laxity Questionnaire (VLQ) | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  7-point Likert-type subjective scale, ranging from very loose to very tight. Scores below 4 (neither loose nor tight) indicate vaginal laxity.
Change in Pain assessed by NRS | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  Pain intensity perceived during the insertion of vaginal dilators of varying diameters (ranging from 20 to 30 mm) will be assessed using the Numeric Rating Scale, where 0 indicates no pain and 10 represents the worst possible pain.
Change in Urinary Symptoms by International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form | Baseline, end of treatment period (5 weeks), and three months post-treatment.
  It is a brief 4-item questionnaire designed to assess the frequency, severity, and impact of urinary incontinence on quality of life.
Change in Health- related quality of Life by SF-12 | Baseline, end of treatment period (6 weeks), and three months post-treatment.
  It consists of 12 items that yield two summary scores: physical and mental components. The response options follow a Likert-type scale that measures either intensity or frequency. Scale scores range from 0 to 100, with 0 indicating the worst health status and 100 the best.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Quezada Bascuñán, Ms, Principal Investigator — University of Castilla-La Mancha; Asunción Ferri Morales, PhD, Study Chair — University of Castilla-La Mancha
Locations (1):
- University of Castilla-La Mancha, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naumova I, Castelo-Branco C. Current treatment options for postmenopausal vaginal atrophy. Int J Womens Health. 2018 Jul 31;10:387-395. doi: 10.2147/IJWH.S158913. eCollection 2018. PMID 30104904
- [Background] Potter N, Panay N. Vaginal lubricants and moisturizers: a review into use, efficacy, and safety. Climacteric. 2021 Feb;24(1):19-24. doi: 10.1080/13697137.2020.1820478. Epub 2020 Sep 29. PMID 32990054
- [Background] Wiegerinck AIP, Thomsen A, Hisdal J, Kalvoy H, Tronstad C. Electrical Impedance Plethysmography Versus Tonometry To Measure the Pulse Wave Velocity in Peripheral Arteries in Young Healthy Volunteers: a Pilot Study. J Electr Bioimpedance. 2021 Dec 30;12(1):169-177. doi: 10.2478/joeb-2021-0020. eCollection 2021 Jan. PMID 35111272
- [Background] Shifren JL, Crandall CJ, Manson JE. Menopausal Hormone Therapy. JAMA. 2019 Jun 25;321(24):2458-2459. doi: 10.1001/jama.2019.5346. No abstract available. PMID 31145419
- [Background] Roy S, Caillouette JC, Roy T, Faden JS. Vaginal pH is similar to follicle-stimulating hormone for menopause diagnosis. Am J Obstet Gynecol. 2004 May;190(5):1272-7. doi: 10.1016/j.ajog.2003.12.015. PMID 15167829
- [Background] undefined
- [Background] Tan O, Bradshaw K, Carr BR. Management of vulvovaginal atrophy-related sexual dysfunction in postmenopausal women: an up-to-date review. Menopause. 2012 Jan;19(1):109-17. doi: 10.1097/gme.0b013e31821f92df. PMID 22011753
- [Background] Sarmento ACA, Costa APF, Vieira-Baptista P, Giraldo PC, Eleuterio J Jr, Goncalves AK. Genitourinary Syndrome of Menopause: Epidemiology, Physiopathology, Clinical Manifestation and Diagnostic. Front Reprod Health. 2021 Nov 15;3:779398. doi: 10.3389/frph.2021.779398. eCollection 2021. PMID 36304000
- [Background] Takahashi TA, Johnson KM. Menopause. Med Clin North Am. 2015 May;99(3):521-34. doi: 10.1016/j.mcna.2015.01.006. PMID 25841598